CLINICAL TRIAL: NCT00584155
Title: Evaluation of Lactated Ringers for Protection From Cisplatin Ototoxicity.
Brief Title: Protection From Cisplatin Ototoxicity by Lactated Ringers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the university.
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Dini Chissoe, Study Coordinator, University of Oklahoma
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Lactated Ringers - Berryhill
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2010-06

CONDITIONS: Hearing Loss
Keywords: Cisplatin Ototoxicity; Lactated Ringer's; Ear Cancer; Hearing loss; Hearing loss due to Cisplatin Ototoxicity
MeSH Terms: conditions — Hearing Loss; Ear Neoplasms | interventions — Saline Solution; Ofloxacin; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Each patient will receive a bottle containing normal saline and 0.03% ofloxacin.
  Interventions: Drug: Normal Saline and 0.3% ofloxacin
- 2 (Experimental): Each patient will receive a bottle containing Lactated Ringer's solution and 0.03% ofloxacin.
  Interventions: Drug: Lactated Ringer's with 0.03% Ofloxacin

INTERVENTIONS:
Drug: Normal Saline and 0.3% ofloxacin — The patient will be instructed to place one dropper full of solution in the external auditory canal. The bottle will be marked right or left ear and are only to be used in the designated ear. The drops will be administered at the start time, 30 minutes after chemotherapy starts and hourly for 4 hours after infusion.
  Arms: 1
Drug: Lactated Ringer's with 0.03% Ofloxacin — The patient will be instructed to place one dropper full of solution in the external auditory canal. The bottle will be marked right or left ear. The drops will be administered at the start time, 30 minutes after chemotherapy starts and hourly for 4 hours after infusion.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if Lactated Ringer's solution is effective in patients undergoing chemotherapy with cisplatin for head and neck cancer in regards to cisplatin-induced hearing loss.

DETAILED DESCRIPTION:
About one-third of people who have been given Cisplatin, as part of their chemotherapy treatment, develop hearing loss. The purpose of this study is to determine if some degree of hearing loss can be prevented by use of Lactated Ringer's solution in the middle ear. To study this, patients will use drops in their ears; Lactated Ringer's will be placed in one ear and an inactive saline solution will be placed in the other. Ofloxacin, an eardrop antibiotic will be placed in each ear at the same time. Each participant will receive a hearing evaluation before each dose of Cisplatin and another evaluation 2 to 4 weeks after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer to be treated with cisplatin.
* Patients expected to receive a minimum of 3 rounds of chemotherapy.
* Patients receiving a minimum dose of cisplatin of 70 mg/m2

Exclusion Criteria:

* Patients who have had middle ear surgery.
* Patients who have active external or middle ear disease
* Patients who have preceding pure tone average of >40 dB HL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pre-treatment audiogram will be compared with the post treatment audiogram. The differences between the two will be calculated and compared to the differences in the opposite ear. | Patients will be enrolled in the study for 4-6 weeks from the initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Berryhill, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States